CLINICAL TRIAL: NCT03706235
Title: Evaluation of the Performance of the Clinical Genomics Colvera Test in the Detection of Disease Recurrence in Patients Diagnosed With Colorectal Cancer- "NOVA"
Brief Title: Colvera for Detection of Disease Recurrence
Acronym: NOVA
Status: Completed | Type: Observational
Sponsor: Clinical Genomics Pathology (Industry)
Responsible Party: Sponsor
Other Study IDs: CG001
Record Dates: First submitted 2018-10-11; First posted 2018-10-15 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Adenocarcinoma
MeSH Terms: interventions — Blood Specimen Collection; Phlebotomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples are used to isolate cf DNA for identification of methylated markers. Leftover plasma with or without extracted DNA may be kept to repeat assays.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No recurrence: Subjects at least 30 days from end of primary treatment for colorectal cancer in a clinically indicated surveillance program (e.g. ASCO, NCCN) provide a blood sample before the next clinically indicated surveillance scan/imaging. Imaging documents no recurrence.
  Interventions: Other: Blood draw (venipuncture)
- Recurrence: Subjects at least 30 days from end of primary treatment for colorectal cancer in a clinically indicated surveillance program (e.g. ASCO, NCCN) provide a blood sample before the next clinically indicated surveillance scan/imaging or imaging has confirmed recurrence. Imaging documents recurrence.
  Interventions: Other: Blood draw (venipuncture)

INTERVENTIONS:
Other: Blood draw (venipuncture) — Draw 40 mls of blood from eligible subjects. Process and ship samples to sponsor.

SUMMARY:
To compare the sensitivity and specificity estimates of Colvera with that of a commercially available CEA test for detection of recurrent disease in CRC subjects who are undergoing surveillance for recurrence.

DETAILED DESCRIPTION:
This is an observational, prospective comparison study, where blood is collected for assay of methylated BCAT1 and IKZF1 DNA and CEA, from subjects who have undergone curative treatment for primary CRC of stages II and III (AJCC) and who are in remission and scheduled for follow-up radiological imaging as part of their surveillance program for recurrence. Participation is for one visit only as part of each subject's surveillance-monitoring schedule. Two K2-EDTA blood tubes and two PAXgene™ tubes will be collected Any evidence of methylated BCAT1 and/or IKZF1 DNA in blood represents a Colvera "positive" result. CEA levels of 5ug/L or higher will represent a "positive" result. Sensitivity and specificity of the Colvera and CEA test will be estimated and compared in a paired fashion in each case where recurrence status has been investigated and determined by the site clinical management team. Blood testing shall be performed and analyzed by qualified staff blinded to clinical status. This is a cross-sectional observational non-significant risk study, and test results will not be used for clinical management, i.e. there will be no interventions in subjects consenting to participate in this Research Study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years or older, and capable and willing to provide informed consent.
2. Subject has undergone curative treatment for primary CRC of stages II and III (AJCC).
3. Subject has no clinical evidence of disease (NED) (after initial treatment)
4. Subject has concluded course of initial treatment for primary CRC (i.e. end of surgery, chemotherapy and/or radiotherapy)
5. Subject is willing/able to provide a blood sample

Exclusion Criteria:

1. Subject has evidence of residual disease.
2. Subject has other organ cancer at the time of recruitment.
3. Subject has prior history of recurrent CRC.
4. Subject has concurrent serious non-neoplastic illness that makes enrollment impractical or clinically inappropriate.
5. Subject is receiving chemo- or radiotherapy at the time of blood collection, or between blood collection and radiological imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects who have undergone curative treatment for primary Colon or rectal cancer of stages II and III (AJCC), and who are in remission and scheduled for clinical follow-up (usually radiological imaging) as part of their surveillance program for recurrence.
Sampling Method: Non-Probability Sample
Enrollment: 488 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive predictive value and negative predictive value | 1.5 years
  on positive or negative Colvera and CEA test results

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Torrance Memorial Physician Network, Redondo Beach, California
  - Bayhealth, Dover, Delaware
  - Rush University Medical Center, Chicago, Illinois
  - NorthShore Health System, Evanston, Illinois
  - Indiana University, Indianapolis, Indiana
  - Colon and Rectal Surgery Associates, Metairie, Louisiana
  - Providence Hospital-Ascension Health, Novi, Michigan
  - Virginia Piper Cancer Institute-Allina Health, Minneapolis, Minnesota
  - Essex Oncology, Belleville, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - University Hospitals, Cleveland, Ohio
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The data collected by recruiting sites is captured without any PHI or identifiers in an Electronic Data Capture system managed for the sponsor by a CRO.
Supporting Information: Study Protocol, SAP, CSR